CLINICAL TRIAL: NCT02611427
Title: Increasing Long-Term Physical Activity After Lumbar Spine Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2015-142
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lumbar Spine Degenerative Changes
Keywords: spine; lumbar; postoperative; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Education/Self-efficacy (Active Comparator): Booklet about physical activity, movement monitoring device, encouragement
  Interventions: Behavioral: Education/Self-efficacy
- Education (Active Comparator): Booklet about physical activity
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education/Self-efficacy — The education/self-efficacy group will 1) receive information about benefits of physical activity and national activity guidelines, 2) receive instruction on how to increase lifestyle walking, 3) use movement monitoring devices, 4) make a walking contract and 5) receive interval contract-directed encouragement from study personnel.
  Arms: Education/Self-efficacy
Behavioral: Education — The education group will receive information about safe physical activity.
  Arms: Education

SUMMARY:
After recuperating from low back surgery patients often perpetuate a sedentary lifestyle because they are concerned about injury and recurrent pain. The objective of this study is to test the feasibility of a program to increase lifestyle walking starting several months after low back surgery.

DETAILED DESCRIPTION:
The primary objective of this RCT is to compare energy expenditure from walking between an experimental group that receives a multi-component intervention based on the Health Belief Model of Behavior Change versus a control group. Patients who had surgery for a degenerative condition will be randomized postop when their surgeons deem them orthopedically stable to increase walking (at about 3 months).

ELIGIBILITY:
* Inclusion Criteria: Patients will be eligible if they had lumbar surgery for a degenerative condition and their surgeon deems it safe for them to walk more.
* Exclusion Criteria: Patients will be excluded if they had any new cardiopulmonary symptoms since surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Weekly energy expenditure in kilocalories per week as measured by the Paffenbarger Physical Activity and Exercise Index | 16 weeks
  Change in enrollment to 16-week Paffenbarger Physical Activity and Exercise Index

SECONDARY OUTCOMES:
Disability due to pain as measured by the Oswestry Disability Index | 16 weeks
  Change in enrollment to 16-week Oswestry Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Choi TN, Westermann H, Wenderoth S, Hollenberg JP, Wells MT, Isen AM, Jobe JB, Allegrante JP, Charlson ME. Increasing physical activity in patients with asthma through positive affect and self-affirmation: a randomized trial. Arch Intern Med. 2012 Feb 27;172(4):337-43. doi: 10.1001/archinternmed.2011.1316. Epub 2012 Jan 23. PMID 22269593
- [Background] Mancuso CA, Perna M, Sargent AB, Salmon JE. Perceptions and measurements of physical activity in patients with systemic lupus erythematosus. Lupus. 2011 Mar;20(3):231-42. doi: 10.1177/0961203310383737. Epub 2010 Dec 23. PMID 21183562
- [Background] Mancuso CA, Cammisa FP, Sama AA, Hughes AP, Ghomrawi HM, Girardi FP. Development and testing of an expectations survey for patients undergoing lumbar spine surgery. J Bone Joint Surg Am. 2013 Oct 2;95(19):1793-800. doi: 10.2106/JBJS.L.00338. PMID 24088972
- [Background] Mancuso CA, Choi TN, Westermann H, Wenderoth S, Wells MT, Charlson ME. Improvement in asthma quality of life in patients enrolled in a prospective study to increase lifestyle physical activity. J Asthma. 2013 Feb;50(1):103-7. doi: 10.3109/02770903.2012.743150. Epub 2012 Nov 22. PMID 23173979
- [Background] Mancuso CA, Duculan R, Stal M, Girardi FP. Patients' expectations of lumbar spine surgery. Eur Spine J. 2015 Nov;24(11):2362-9. doi: 10.1007/s00586-014-3597-z. Epub 2014 Oct 8. PMID 25291976